CLINICAL TRIAL: NCT00334126
Title: A Randomized, Double-blind, Placebo-controlled, Parallel Group Study to Evaluate the Efficacy and Safety of Paliperidone ER Compared to Quetiapine in Subjects With an Acute Exacerbation of Schizophrenia
Brief Title: Evaluation of Effectiveness and Safety of Paliperidone ER (Extended-release) Compared With Quetiapine in Patients With Schizophrenia
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Johnson & Johnson Pharmaceutical Research & Development, L.L.C. (Industry)
Collaborators: Janssen, LP (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CR010501
Record Dates: First submitted 2006-06-02; First posted 2006-06-06 (Estimated); Last update posted 2011-05-18 (Estimated); Status verified 2010-03

CONDITIONS: Schizophrenia
Keywords: Schizophrenia; Antipsychotic; paliperidone; quetiapine; Seroquel; placebo
MeSH Terms: conditions — Schizophrenia

INTERVENTIONS:
Drug: paliperidone ER tablets, quetiapine tablets, placebo - all over encapsulated

SUMMARY:
The purpose of this study is to evaluate the efficacy (effectiveness of drug) and safety of the antipsychotic paliperidone ER compared to another antipsychotic, quetiapine, and to placebo in patients who are acutely ill with symptoms of schizophrenia.

DETAILED DESCRIPTION:
This is a randomized (patients are assigned different treatments based on chance), double blind (neither the patient nor the physician knows whether drug or placebo is being taken, or at what dosage), placebo controlled, parallel group study to compare the efficacy and safety of paliperidone ER with quetiapine in the treatment of patients who have schizophrenia and are acutely ill. The duration of the study is 42 days. During the first phase (Day 0 - Day 14) patients receive increasing doses of the treatment to which they are assigned (starting with 3mg and increasing to 9 mg or 12 mg of paliperidone ER; starting with 50 mg and increasing to 600 mg or 800 mg of quetiapine; or the same number of capsules of placebo). During the second phase (Day 15 - Day 42), patients continue to take the dose of medication they received on day 14, but may also receive other medications if the investigator determines they are needed to treat ongoing symptoms. The hypothesis of the study is that paliperidone ER is better than quetiapine in the short term for treating acutely ill patients with schizophrenia. Primary outcome is change on the total score of the PANSS (Positive and Negative Syndrome scale for Schizophrenia) in the first phase of the study (Day 0 - Day 14). Secondary outcomes include time to response, time to readiness for discharge, and additional medication use in the second phase of the study (Day 15- Day 42) for patients receiving paliperidone ER compared to quetiapine. Safety of paliperidone ER compared with quetiapine throughout the study (Day 0 - Day 42) will be based on reported adverse events, results of laboratory tests (hematology, biochemistry, and urinalysis), vital signs (blood pressure, pulse, and weight), electrocardiogram, and movement disorder scales (Abnormal Involuntary Movement Scale, Barnes Akathisia Scale, and Simpson-Angus Rating Scale). Patients may participate in a pharmacogenomic (DNA) analysis, if they choose to do so. Patients receive study drug by mouth for a total of 42 days. Study medications will be increased to maximum tolerated doses of Paliperidone ER 9mg or 12mg/day and Quetiapine 600mg or 800mg at day 8. From day 15 through day 42 (end of study) all patients will be eligible for additional psychotropic medications at investigators' discretion.

ELIGIBILITY:
Inclusion Criteria:

* Diagnostic and Statistical Manual - Fourth Edition (DSM-IV) diagnosis of schizophrenia (paranoid, disorganized or undifferentiated type)
* score of >=4 on at least two of a subset of selected PANSS items and a total score on these five items of >=17
* score of >=5 on the CGI-S (clinical global impression - severity)
* body weight of at least 60kg and willing to be hospitalized for 9 days initially

Exclusion Criteria:

* A primary active mental illness diagnosis other than schizophrenia
* subjects whose psychotic symptoms can be explained by substance intake or medical illness
* pregnancy, breast-feeding, or planning to become pregnant
* a history of treatment resistance (defined by failure to respond to 2 adequate trials of different antipsychotic medications or clozapine given at adequate dose for sufficient time)
* unstable or significant medical illness that would increase risk of taking study medication or would confuse the interpretation of the study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 399 (Actual)
Dates: Start 2006-04; Study Completion 2007-09 (Actual)

PRIMARY OUTCOMES:
Reduction in total PANSS ( Positive and Negative Syndrome Scale) from baseline to endpoint at Day 14

SECONDARY OUTCOMES:
Time to response (based on reduction in PANSS plus Clinical Global Impression - Change) and readiness for discharge, utilization of health care resources and polypharmacy use in patients receiving paliperidone ER or quetiapine

CONTACTS AND LOCATIONS:
Overall Officials: Johnson & Johnson Pharmaceutical Research & Development, L.L. C. Clinical Trial, Study Director — Johnson & Johnson Pharmaceutical Research & Development, L.L.C.

REFERENCES:
- [Derived] Canuso CM, Dirks B, Carothers J, Kosik-Gonzalez C, Bossie CA, Zhu Y, Damaraju CV, Kalali AH, Mahmoud R. Randomized, double-blind, placebo-controlled study of paliperidone extended-release and quetiapine in inpatients with recently exacerbated schizophrenia. Am J Psychiatry. 2009 Jun;166(6):691-701. doi: 10.1176/appi.ajp.2009.08040613. Epub 2009 May 1. PMID 19411369
- See also: A randomized, double blind, placebo-controlled, parallel group study to evaluate the efficacy and safety of paliperidone ER compared to quetiapine in subjects with an acute exacerbation schizophrenia — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_JNJ_6051&studyid=715&filename=CR010501_CSR.pdf